CLINICAL TRIAL: NCT03771469
Title: Validation of Sleep Questionnaires in the Down Syndrome Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Derek Lam, MD, MPH, Assistant Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00018522
Record Dates: First submitted 2018-08-10; First posted 2018-12-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea; Down Syndrome
Keywords: OSA; obstructive sleep apnea; Down syndrome; sleep questionnaires; sleep study
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome

STUDY DESIGN:
Intervention Model Description: This will be a prospective validation study of a sample of consecutive pediatric Down syndrome patients who are seen through the weekly Down syndrome clinic at OHSU/Doernbecher's.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Questionnaires and sleep studies (Experimental): Caregivers of patients meeting eligibility criteria will be invited to participate. If they agree to participate, baseline SRBD-PSQ, OSA-18, and PedsQL questionnaires along with written informed consent forms will be mailed to them along with their standard scheduling paperwork. Caregivers will be asked to review the consent form and complete the questionnaires and bring the paperwork to clinic on the day of their visit. Sleep study testing will also be ordered prior to their visit so that it can be scheduled within a month of the initial clinic visit and again three months later.
  Interventions: Other: Sleep study

INTERVENTIONS:
Other: Sleep study — Sleep study
  Other Names: polysomnography

SUMMARY:
This will be a prospective validation study of a sample of consecutive pediatric Down syndrome patients who are seen through the weekly Down syndrome clinic at OHSU/Doernbecher's. Questionnaires will be administered to approximately 5 new patients per month. Since this population has a higher prevalence of OSA than the general pediatric population, and OSA is a potentially modifiable determinant of quality of life, validated instruments are critical in assessing disease burden and response to treatment.

DETAILED DESCRIPTION:
Specific Aims:

1. Demonstrate the criterion validity of the Sleep-Related Breathing Disorder subscale of the PSQ as a screening tool for the diagnosis of OSA in children with Down Syndrome, using polysomnography as the gold standard.

   Hypothesis: Compared to the published threshold for a positive screen in the general pediatric population (≥ 7 of 22 positive responses), the threshold for a positive screen that corresponds to an optimal sensitivity and specificity in the Down syndrome population will be significantly different.
2. Demonstrate the construct validity of the OSA-18 as a scale to assess sleep-related quality of life in children with Down Syndrome by comparing OSA-18 scores to an objective measure of disease burden (polysomnography) and a generic quality of life instrument (the Pediatric Quality of Life inventory, PedsQL).

Hypothesis: OSA-18 scores will be significantly associated with the Apnea-Hypopnea Index assessed by polysomnography and the PedsQL Total Score, Physical Health, and Psychosocial Health summary scores.

Background:

1. Obstructive Sleep Apnea and Down Syndrome: Obstructive sleep apnea (OSA) affects 1-5% of children in the US and has been associated with a myriad of health consequences including cardiovascular complications, behavioral disturbances, and neurocognitive dysfunction. In contrast, there is a reported OSA prevalence of 31-79% in children with Down Syndrome due to traits that predispose to OSA including hypotonia, obesity, and craniofacial anatomy such as midfacial and mandibular hypoplasia which can lead to pharyngeal crowding. With increased risk of congenital cardiovascular defects in the Down Syndrome population, it is possible that these children are also at risk of the most serious complications of OSA including pulmonary hypertension.

   OSA has also been shown to have a significant impact on quality of life. Behavioral problems associated with OSA include reduced attention, hyperactivity, irritability and problems with peers. Previous studies in the general pediatric population have shown similar quality of life scores in children with symptoms of OSA as children with asthma and rheumatoid arthritis. In children with Down syndrome, reduced sleep has been associated with reduced cognitive function, memory, poor communication skills, and poor self-help skills. Furthermore, parents of children with sleep disordered breathing often suffer from sleep deprivation themselves which can result in negative impacts on family life, decreased ability to care for their children and higher levels of maternal stress.
2. Subjective Measures of Sleep Disordered Breathing and Obstructive Sleep Apnea: Overnight polysomnography (PSG) is the gold standard for diagnosing OSA in children. However, due to cost and inconvenience, only a minority of patients being evaluated for OSA undergo PSG prior to adenotonsillectomy. One survey study conducted among pediatric otolaryngologists showed that 31% of respondents said they referred children suspected of OSA for PSG "rarely" or "never." In a separate study, 75% of pediatric otolaryngologists surveyed referred for PSG in less than 10% of children with suspected OSA. Commonly cited factors for this include cost of obtaining PSG and delay in obtaining PSG due to availability. In addition, a substantial proportion of patients referred for PSG are either lost to follow-up or experience significant delays in treatment due to testing. As a result, alternative methods of screening for or diagnosing OSA have been explored that are cheaper and less burdensome. This includes a variety of questionnaires that were designed to screen the pediatric population for symptoms of sleep disordered-breathing (SDB) and assess its impact on quality of life within a clinic setting. The Sleep-Related Breathing Disorders subscale of the Pediatric Sleep Questionnaire (SRBD-PSQ) was developed to screen for SDB using 3 categories: daytime sleepiness, snoring, and behavioral disturbances.3 This has previously been validated in children aged 2-18 within the general pediatric population. The OSA-18 is a survey that measures the impact of SDB or OSA on disease-specific quality of life in children by assessing common manifestations of the disease including sleep disturbance, emotional distress, daytime function, and caregiver concerns. This questionnaire has been validated in children ages 6 months to 12 years. Validated subjective measures like these capture different aspects of the disease experience than objective measures like PSG. They can also be used to assess large numbers of patients with far less burden and expense than PSG which frequently has long wait times due to limited capacity.
3. No Validated Screening instruments or OSA-related QOL measures in Down Syndrome: Despite the high prevalence of OSA in the Down syndrome population and the availability of widely used questionnaires for SDB, screening for SDB is generally inconsistent in this population. Even when parental report of symptoms of SDB is solicited, multiple studies have demonstrated poor diagnostic accuracy of parental history compared to PSG. A recent study investigating parental assessment of the symptoms of SDB found that 66% of Down syndrome patients had frequent symptoms consistent with SDB including snoring, witnessed apnea, and restless sleep. However, there was no association between the frequency of these symptoms and diagnosis with OSA. Other studies have similarly demonstrated poor diagnostic accuracy of parental history with respect to PSG findings. For this reason, the most recent American Academy of Pediatrics (AAP) guideline regarding management of Down syndrome patients has recommended routine screening for OSA using PSG in all patients by the age of 4, regardless of symptomatology. There are currently no validated instruments for screening for OSA or assessing OSA-related quality of life in the Down syndrome population.

ELIGIBILITY:
Inclusion Criteria:

Children with Down syndrome aged 2-17 years who are seen through the Down syndrome clinic at Oregon Health and Science University who either have a recently completed sleep study (within the past 6 months and no surgical treatment for OSA since then) or who will be having a sleep study.

Exclusion Criteria:

* Presence of tracheostomy
* Presence of subglottic or tracheal stenosis
* Severe cardiopulmonary disease requiring supplemental oxygen
* Parents or caregivers who are unable to read written English or Spanish

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) from polysomnography | AHI collected at initial sleep study and 3 months later (if a second sleep study is needed as determined by doctor)
  Overnight attended polysomnography is the gold standard for diagnosis of OSA. Assessment of sleep staging is done through electroencephalogram, electro-oculogram, and submental electromyogram. The primary output parameter that is commonly used to diagnose and characterize the severity of OSA is the apnea-hypopnea index (AHI).

SECONDARY OUTCOMES:
Sleep Related Breathing Disorder subscale total of the Pediatric Sleep Questionnaire (SRBD-PSQ) | SRBD score tallied at initial clinic visit.
  The SRBD-PSQ is a subjective instrument with 22-items that was designed to screen for sleep-related disordered breathing in the general pediatric population. Each question is answered with a yes (1 point), no (0 points), or don't know (0 points). The total number of points is added up, and that sum is divided by the number of questions answered to produce a ratio. When assessing the ratio, a figure greater than 0.3 is considered a positive screening for OSA. There are no subscales on this questionnaire.
Sleep-Related Quality of Life (OSA-18 total score) | OSA-18 total collected at initial clinic visit.
  The OSA-18 is a subjective measure of disease-specific quality of life survey for sleep disordered breathing. It contains 18 questions. These questions are scored on a 7 point Likert scale, with "1" being the worst outcome and "7" being the best outcome. These numeric scores are totaled to produce one overall sum, with a range from 7 to 126.
Generic Quality of Life | PedsQL summary scores collected at initial clinic visit.
  The Pediatric Quality of Life Inventory (PedsQL) is a validated generic quality of life measure encompassing 4 multidimensional scales (Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning) with three Summary Scores (Total Score, Physical Health Summary Score, Psychosocial Health Summary Score). The number of questions varies by age group but falls within 20-25 questions. The questions use 5-point Likert scale from 0 (Never) to 4 (Almost always). Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0.). Dimensions are scored by transforming into mean score = Sum of the items over the number of items answered. For each of the 4 scales, higher scores indicate better HRQOL (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Derek Lam, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Doernbecher Children's Hospital, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Only the PI and members of the study team will have direct access to identifiable private information. Subjects will be assigned a unique randomly generated study identification number and extracted datasets will be coded for use in subsequent analysis.

REFERENCES:
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Goffinski A, Stanley MA, Shepherd N, Duvall N, Jenkinson SB, Davis C, Bull MJ, Roper RJ. Obstructive sleep apnea in young infants with Down syndrome evaluated in a Down syndrome specialty clinic. Am J Med Genet A. 2015 Feb;167A(2):324-30. doi: 10.1002/ajmg.a.36903. Epub 2015 Jan 13. PMID 25604659
- [Background] de Miguel-Diez J, Villa-Asensi JR, Alvarez-Sala JL. Prevalence of sleep-disordered breathing in children with Down syndrome: polygraphic findings in 108 children. Sleep. 2003 Dec 15;26(8):1006-9. doi: 10.1093/sleep/26.8.1006. PMID 14746382
- [Background] Maris M, Verhulst S, Wojciechowski M, Van de Heyning P, Boudewyns A. Prevalence of Obstructive Sleep Apnea in Children with Down Syndrome. Sleep. 2016 Mar 1;39(3):699-704. doi: 10.5665/sleep.5554. PMID 26612391
- [Background] Baldassari CM, Mitchell RB, Schubert C, Rudnick EF. Pediatric obstructive sleep apnea and quality of life: a meta-analysis. Otolaryngol Head Neck Surg. 2008 Mar;138(3):265-273. doi: 10.1016/j.otohns.2007.11.003. PMID 18312869
- [Background] Quine L. Sleep problems in children with mental handicap. J Ment Defic Res. 1991 Aug;35 ( Pt 4):269-90. doi: 10.1111/j.1365-2788.1991.tb00402.x. PMID 1757978
- [Background] Breslin J, Spano G, Bootzin R, Anand P, Nadel L, Edgin J. Obstructive sleep apnea syndrome and cognition in Down syndrome. Dev Med Child Neurol. 2014 Jul;56(7):657-64. doi: 10.1111/dmcn.12376. Epub 2014 Jan 29. PMID 24471822
- [Background] Carter M, McCaughey E, Annaz D, Hill CM. Sleep problems in a Down syndrome population. Arch Dis Child. 2009 Apr;94(4):308-10. doi: 10.1136/adc.2008.146845. Epub 2008 Sep 11. PMID 18786953
- [Background] Huang YS, Guilleminault C, Li HY, Yang CM, Wu YY, Chen NH. Attention-deficit/hyperactivity disorder with obstructive sleep apnea: a treatment outcome study. Sleep Med. 2007 Jan;8(1):18-30. doi: 10.1016/j.sleep.2006.05.016. Epub 2006 Dec 6. PMID 17157069
- [Background] Mitchell RB, Kelly J. Behavior, neurocognition and quality-of-life in children with sleep-disordered breathing. Int J Pediatr Otorhinolaryngol. 2006 Mar;70(3):395-406. doi: 10.1016/j.ijporl.2005.10.020. PMID 16321451
- [Background] Friedman NR, Perkins JN, McNair B, Mitchell RB. Current practice patterns for sleep-disordered breathing in children. Laryngoscope. 2013 Apr;123(4):1055-8. doi: 10.1002/lary.23709. Epub 2013 Feb 4. PMID 23382017
- [Background] Mitchell RB, Pereira KD, Friedman NR. Sleep-disordered breathing in children: survey of current practice. Laryngoscope. 2006 Jun;116(6):956-8. doi: 10.1097/01.MLG.0000216413.22408.FD. PMID 16735907
- [Background] Boss EF, Benke JR, Tunkel DE, Ishman SL, Bridges JF, Kim JM. Public insurance and timing of polysomnography and surgical care for children with sleep-disordered breathing. JAMA Otolaryngol Head Neck Surg. 2015 Feb;141(2):106-11. doi: 10.1001/jamaoto.2014.3085. PMID 25503255
- [Background] Santoro SL, Yin H, Hopkin RJ. Adherence to Symptom-Based Care Guidelines for Down Syndrome. Clin Pediatr (Phila). 2017 Feb;56(2):150-156. doi: 10.1177/0009922816652416. Epub 2016 Jul 19. PMID 27260508
- [Background] Friedman NR, Ruiz AG, Gao D, Ingram DG. Accuracy of Parental Perception of Nighttime Breathing in Children with Down Syndrome. Otolaryngol Head Neck Surg. 2018 Feb;158(2):364-367. doi: 10.1177/0194599817726286. Epub 2017 Sep 5. PMID 28871845
- [Background] Nehme J, LaBerge R, Pothos M, Barrowman N, Hoey L, Monsour A, Kukko M, Katz SL. Predicting the presence of sleep-disordered breathing in children with Down syndrome. Sleep Med. 2017 Aug;36:104-108. doi: 10.1016/j.sleep.2017.03.032. Epub 2017 May 31. PMID 28735906
- [Background] Ng DK, Chan CH, Cheung JM. Children with Down syndrome and OSA do not necessarily snore. Arch Dis Child. 2007 Nov;92(11):1047-8. No abstract available. PMID 17954492
- [Background] Shott SR, Amin R, Chini B, Heubi C, Hotze S, Akers R. Obstructive sleep apnea: Should all children with Down syndrome be tested? Arch Otolaryngol Head Neck Surg. 2006 Apr;132(4):432-6. doi: 10.1001/archotol.132.4.432. PMID 16618913
- [Background] Lin SC, Davey MJ, Horne RS, Nixon GM. Screening for obstructive sleep apnea in children with Down syndrome. J Pediatr. 2014 Jul;165(1):117-22. doi: 10.1016/j.jpeds.2014.02.032. Epub 2014 Mar 25. PMID 24679609
- [Background] Bull MJ; Committee on Genetics. Health supervision for children with Down syndrome. Pediatrics. 2011 Aug;128(2):393-406. doi: 10.1542/peds.2011-1605. Epub 2011 Jul 25. PMID 21788214
- [Background] Spruyt K, Gozal D. Pediatric sleep questionnaires as diagnostic or epidemiological tools: a review of currently available instruments. Sleep Med Rev. 2011 Feb;15(1):19-32. doi: 10.1016/j.smrv.2010.07.005. Epub 2010 Oct 8. PMID 20934896
- [Background] Skotko BG, Macklin EA, Muselli M, Voelz L, McDonough ME, Davidson E, Allareddy V, Jayaratne YS, Bruun R, Ching N, Weintraub G, Gozal D, Rosen D. A predictive model for obstructive sleep apnea and Down syndrome. Am J Med Genet A. 2017 Apr;173(4):889-896. doi: 10.1002/ajmg.a.38137. Epub 2017 Jan 26. PMID 28124477
- [Background] Chervin RD, Weatherly RA, Garetz SL, Ruzicka DL, Giordani BJ, Hodges EK, Dillon JE, Guire KE. Pediatric sleep questionnaire: prediction of sleep apnea and outcomes. Arch Otolaryngol Head Neck Surg. 2007 Mar;133(3):216-22. doi: 10.1001/archotol.133.3.216. PMID 17372077
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Franco RA Jr, Rosenfeld RM, Rao M. First place--resident clinical science award 1999. Quality of life for children with obstructive sleep apnea. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):9-16. doi: 10.1067/mhn.2000.105254. PMID 10889473
- [Background] Goldstein NA, Fatima M, Campbell TF, Rosenfeld RM. Child behavior and quality of life before and after tonsillectomy and adenoidectomy. Arch Otolaryngol Head Neck Surg. 2002 Jul;128(7):770-5. doi: 10.1001/archotol.128.7.770. PMID 12117332
- [Background] Sohn H, Rosenfeld RM. Evaluation of sleep-disordered breathing in children. Otolaryngol Head Neck Surg. 2003 Mar;128(3):344-52. doi: 10.1067/mhn.2003.4. PMID 12646836
- [Background] Mitchell RB, Kelly J, Call E, Yao N. Long-term changes in quality of life after surgery for pediatric obstructive sleep apnea. Arch Otolaryngol Head Neck Surg. 2004 Apr;130(4):409-12. doi: 10.1001/archotol.130.4.409. PMID 15096422
- [Background] Mitchell RB, Kelly J. Quality of life after adenotonsillectomy for SDB in children. Otolaryngol Head Neck Surg. 2005 Oct;133(4):569-72. doi: 10.1016/j.otohns.2005.05.040. PMID 16213931
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Marcus CL, Keens TG, Bautista DB, von Pechmann WS, Ward SL. Obstructive sleep apnea in children with Down syndrome. Pediatrics. 1991 Jul;88(1):132-9. PMID 1829151